CLINICAL TRIAL: NCT00606294
Title: A Study Using Fluorine-18-Labeled Fluoro-Misonidazole Positron Emission Tomography To Detect Hypoxia in Head and Neck Cancer Patients
Brief Title: Using Fluorine-18-Labeled Fluoro-Misonidazole Positron Emission Tomography To Detect Hypoxia in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-070
Record Dates: First submitted 2008-01-10; First posted 2008-02-01 (Estimated); Results first posted 2020-07-10 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: Head; Neck; 04-070
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — fluoromisonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (closed to accrual) (Experimental): Cohort 1 (closed to accrual) Cohort 1 (closed to accrual) There will be no change or intervention in a patient's treatment regime using chemoradiation where both the primary and the neck nodes receive 70Gy. This is currently one accepted standard of care. In a subcohort of patients in Cohort 1 with tumors that are positive for HPV who exhibited no evidence of hypoxia on their baseline 18F-FMISO PET/ CT scan or whose tumors have early resolution of hypoxia on their repeat early response 18F-FMISO PET/CT scan will undergo an alternative treatment where the primary tumor site receives 70Gy while the neck nodes receive 60Gy followed by a planned FDG PET/CT scan and observation.
  Interventions: Radiation: fluorine-18-labeled fluoro-misonidazole (18F-FMISO); Device: 18F-FMISO PET scan; Device: MRI; Device: FDG PET/CT scan
- Cohort 2 (closed to accrual) (Experimental): Experimental: Cohort 2 (closed to accrual) Cohort 2 HPV+ tumors that demonstrate no evidence of hypoxia on an 18F-FMISO PET scan will receive 30Gy to the surgical bed and neck lymph nodes concurrent with standard chemotherapy followed by a 3-4 month post-treatment neck dissection. In patients who exhibit a complete response with this method of treatment, no further treatment is necessary. For patients within this select group who still have pathologic nodal disease, further standard chemoradiation will be given. All other patients in this cohort (i.e. those who are not in the select HPV+ tumor group outlined above) will receive standard of care treatment following their surgery.
  Interventions: Radiation: fluorine-18-labeled fluoro-misonidazole (18F-FMISO); Device: 18F-FMISO PET scan; Device: MRI; Device: FDG PET/CT scan

INTERVENTIONS:
Radiation: fluorine-18-labeled fluoro-misonidazole (18F-FMISO)
Device: 18F-FMISO PET scan
Device: MRI
Device: FDG PET/CT scan

SUMMARY:
The main purpose of this study is to evaluate low oxygen areas called hypoxia within tumors. These low oxygen areas are thought to be the reason why tumors are more resistant to chemotherapy and radiation treatment.

An imaging technique using a hypoxia tracer called fluoromisonidazole (FMISO) can detect low oxygen areas within a tumor. This imaging technique, called a PET scan, uses positively charged particles to detect slight changes in the body's biochemistry and metabolism. FMISO PET scans have been performed in patients with head and neck cancer and have shown the ability to detect low oxygen areas within tumors.

ELIGIBILITY:
Inclusion Criteria for Cohort 1 and Cohort 2 :

* Histologically confirmed diagnosis of head and neck carcinoma (excluding nasopharynx, paranasal sinus, salivary, and thyroid malignancies)Any unknown primary squamous cell carcinoma of head and neck with gross nodes is allowed (2002 AJCC)
* 18 years of age or older
* Must not have received prior radiation therapy or chemotherapy for this diagnosis. Patients who have had their primary site tumor removed by surgery but still present with grossly enlarged lymph nodes are eligible for this study.
* Karnofsky performance status ≥ 70.

Exclusion Criteria for Cohort 1 and Cohort 2:

* all nasopharyngeal, paranasal sinus, salivary cancer, and thyroid malignancies
* prior chemotherapy or radiotherapy within the last three years
* patients that underwent previous surgical resection for the same disease (except for biopsy or surgery removing primary site tumor but still present with grossly enlarged lymph nodes)
* any prior radiotherapy to the head and neck region
* pregnant (confirmed by serum b-HCG in women of reproductive age) or breast feeding

Subject Exclusion Criteria for Optional Contrast MRIs

• Subjects with a known contraindication to the standard MRI contrast agent (Gadavist, a gadolinium-based contrast agent) and/or a recent estimated glomerular filtration rate (eGFR) of 30 or less will be excluded from all DCE-MRIs, and will instead receive non-contrast MRIs at the DCE-MRI time points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2 (Closed to Accrual): Cohort 2 (closed to accrual) Cohort 2 HPV+ tumors that demonstrate no evidence of hypoxia on an 18F-FMISO PET scan will receive 30Gy to the surgical bed and neck lymph nodes concurrent with standard chemotherapy followed by a 3-4 month post-treatment neck dissection. In patients who exhibit a complete response with this method of treatment, no further treatment is necessary. For patients within this select group who still have pathologic nodal disease, further standard chemoradiation will be given. All other patients in this cohort (i.e. those who are not in the select HPV+ tumor group outlined above) will receive standard of care treatment following their surgery.
Period: Overall Study
Arm/Group | Cohort 1 (Closed to Accrual) | Cohort 2 (Closed to Accrual)
Started | 197 | 19
Completed | 161 | 19
Not Completed | 36 | 0
Not completed — Withdrawal by Subject | 36 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Closed to Accrual) | Cohort 2 (Closed to Accrual) | Total
Number analyzed (Participants) | 197 | 19 | 216
Age, Continuous [Median (Full Range); unit: years] | 58 [25 to 85] | 57 [45 to 70] | 58 [25 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 3 | 26
  Male | 174 | 16 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 9
  Not Hispanic or Latino | 189 | 18 | 207
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 0 | 10
  White | 166 | 17 | 183
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 2 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 197 | 19 | 216

OUTCOME MEASURES:

1. Primary Outcome: To Report Positive Versus Negative Hypoxia Among Head and Neck Cancers Using 18F-FMISO Dynamic PET
Description: For Cohort 1
Time Frame: 4 months
Population: This objective is for Cohort 1 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Closed to Accrual) | Cohort 2 (Closed to Accrual)
Number analyzed (Participants) | 197 | 0
Participants
  Participants who are hypoxia positive | 135 | 0
  Participants who are hypoxia negative | 26 | 0
  Participants declined scans | 36 | 0

2. Primary Outcome: To Determine the Pathologic Complete Response of Low Risk HPV+ Oropharyngeal Cancer Patients Without Hypoxia on 18F-FMISO PET Who Received 30Gy
Description: For Cohort 2 - Feasibility will be determined by the pathologic response rate at time of neck dissection
Time Frame: 4 months
Population: This objective is for Cohort 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Closed to Accrual) | Cohort 2 (Closed to Accrual)
Number analyzed (Participants) | 0 | 19
Participants
  Cohort 2 Pts with a Pathologic Complete Response | 0 | 11
  Cohort 2 Pts w/out a PathologicComplete Response | 0 | 4
  Cohort 2 Participants who were not scanned | 0 | 4

3. Primary Outcome: Improve the Accuracy of Hypoxia Imaging for Head and Neck Cancers Through Pixel by Pixel Kinetic Analysis of 18F-FMISO Tracer of Dynamic PET Images
Description: Cohort 2
Time Frame: At baseline
Population: This objective is for Cohort 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Closed to Accrual) | Cohort 2 (Closed to Accrual)
Number analyzed (Participants) | 0 | 19
Participants
  Cohort 2 Pts Negative at Baseline | 0 | 6
  Cohort 2 Pts Positive at Baseline at Repeat Scan | 0 | 3
  Cohort 2 Pts Negative at Baseline at Repeat Scan | 0 | 9
  Cohort 2 Pts positive at Baseline/withdrew consent | 0 | 1

4. Secondary Outcome: To Detect on Repeat 18F-FMISO PET/CT Scans Whether There is a Reduction of the FMISO-avid or GTVh 5 to 10 Days Into Treatment With Standard Chemoradiotherapy for a Series of Locally Advanced Head and Neck Cancers.
Description: For Cohort 1
Time Frame: 2 weeks from time of scan
Population: N/A - data were not collected
Arm/Group | Cohort 1 (Closed to Accrual) | Cohort 2 (Closed to Accrual)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cohort 1 (Closed to Accrual) | Cohort 2 (Closed to Accrual)
All-Cause Mortality (participants affected / at risk) | 47/197 | 2/19
Serious Adverse Events (participants affected / at risk) | 0/197 | 0/19
Other Adverse Events (participants affected / at risk) | 0/197 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT00606294/Prot_SAP_000.pdf